CLINICAL TRIAL: NCT03721965
Title: An Open-Label, Single-Arm, Phase 1/2 Study Evaluating the Safety and Efficacy of Itacitinib in Combination With Corticosteroids for the Treatment of Steroid-Naive Acute Graft-Versus-Host Disease in Pediatric Subjects
Brief Title: Safety and Efficacy of Itacitinib in Combination With Corticosteroids for Treatment of Graft-Versus-Host Disease in Pediatric Subjects
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to insufficient efficacy in a separate phase III study
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-120; 2018-002253-30 (EudraCT Number)
Expanded Access: NCT03906318 (No longer available)
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Acute Graft-versus-host Disease
Keywords: Acute graft-versus-host disease; GVHD; pediatric; JAK1 inhibitor; corticosteroids
MeSH Terms: interventions — itacitinib; INCB039110; Adrenal Cortex Hormones; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Itacitinib + Corticosteroids (Experimental)
  Interventions: Drug: Itacitinib; Drug: Corticosteroids

INTERVENTIONS:
Drug: Itacitinib — Phase 1: Itacitinib administered orally once daily at the protocol-defined dose according to age cohort, with dose reductions or modifications based on safety assessments. Phase 2: Itacitinib administered orally once daily at the recommended dose from Phase 1.
  Other Names: INCB039110
Drug: Corticosteroids — Phase 1 and 2: Methylprednisolone 2 mg/kg IV daily (or prednisone equivalent) or at a dose that is appropriate for the severity of disease as outlined per local treatment guidelines as background treatment.
  Other Names: prednisone, methylprednisolone

SUMMARY:
The purpose of this study is to evaluate itacitinib in combination with corticosteroids for the treatment of Grades II to IV acute graft-versus-host disease (aGVHD) in steroid-naive pediatric participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants: 12 to < 18 years old (Cohort 1), 6 to < 12 years old (Cohort 2), 2 to < 6 years old (Cohort 3), Weighing > 8 kg to < 2 years old (Cohort 4), and 28 days old to weighing ≤ 8 kg (Cohort 5).
* Undergone 1 allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor and source for hematological malignancies or disorders. Recipients of myeloablative and reduced-intensity conditioning regimens are eligible.
* Clinically suspected Grade II to IV aGVHD as per Mount Sinai Acute GVHD International Consortium (MAGIC) criteria, occurring after allo-HSCT and any GVHD prophylactic medication.
* Evidence of myeloid engraftment.

Exclusion Criteria:

* More than 1 allo-HSCT.
* Received more than 2 days of systemic corticosteroids for aGVHD before the first study drug administration.
* Presence of GVHD overlap syndrome.
* Presence of an active uncontrolled infection.
* Known HIV infection.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection that requires treatment or at risk for HBV reactivation.
* Evidence of relapsed primary disease or have been treated for relapse after the allo-HSCT was performed.
* Any corticosteroid therapy for indications other than GVHD at doses > 1 mg/kg once daily of methylprednisolone (or equivalent) within 7 days of the first study drug administration.
* Receipt of live (including attenuated) vaccines or anticipation of need for such vaccines during the study.
* Receipt of JAK inhibitor therapy after allo-HSCT for any indication.
* Treatment with any other investigational agent, device, or procedure within 21 days (or 5 half-lives, whichever is greater) of enrollment.

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Morariu-Zamfir, MD, Study Director — Incyte Corporation
Locations (37):
- United States (14):
  - City of Hope National Medical Center, Duarte, California
  - Childrens Hospital of Orange County, Orange, California
  - Children's Hospital Colorado - Center for Cancer and Blood Disorders, Aurora, Colorado
  - Nemours/A.I. duPont Hospital for Children, Wilmington, Delaware
  - Nicklaus Children's Hospital, Miami, Florida
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Doernbecher Children's Hospital - Division of Pediatric Hematology, Portland, Oregon
  - Children's Hospital of Philadelphia - Center for Childhood Cancer Research, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- France (7):
  - Centre Hospitalier Universitaire de Rennes, Rennes, Cedex 2
  - Hopitaux Universitaires De Strasbourg, Strasbourg, Cedex
  - CHU de Grenoble, Grenoble
  - Robert Debre Hospital, Paris
  - Hopitaux Universitaires De Strasbourg, Strasbourg
  - CHRU Nancy, Vandœuvre-lès-Nancy
  - CHU Nancy, Vandœuvre-lès-Nancy
- Germany (2):
  - Universitaetsklinikum Aachen, AoeR, Aachen
  - Universitatsklinikum Jena, Klinik fur Kinder und Jugendmedizin, Jena
- Italy (5):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliero Unversitatia Policlinico - Vittorio Emanuele - Presido Ospedaliero G. Rodolico, Catania
  - Fondazione MBBM, Monza
  - Ospedale Pediatrico Bambino Gesu, Roma
  - AOU Citta della Salute e della Scienza di Torino - Ospedale Regina Margherita, Torino
- Spain (3):
  - Hospital Vall D Hebron, Barcelona
  - Hospital Clinico de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (6):
  - Birmingham Childrens Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Great Ormond Street Hospital for Children, London
  - Central Manchester University Hospital - Royal Manchester Children's Hospital, Manchester
  - Royal Marsden Hospital - Surrey, Surrey Quays

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A study of itacitinib in combination with corticosteroids for the treatment of Grades II to IV acute graft-versus-host disease (aGVHD) in pediatric participants 28 days to < 18 years old who were naïve to corticosteroids. The study was conducted from 31-Dec-2019 to 17-Feb-2020.
Pre-assignment Details: A total of 2 participants were screened and included in the study.
Groups:
- Cohort 1 : Itacitinib + Corticosteroids: Itacitinib was administered once a day orally in combination with corticosteroids as per local treatment guidelines.
Period: Overall Study
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Study Terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (2.12) [lower limit 2.12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an AE that began or worsened from Baseline after the first administration of study drug.
Time Frame: up to 45 days
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 2
Participants | 2

2. Primary Outcome: Phase 1: Cmax of Itacitinib When Administered With Corticosteroids
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Day 1: 1, 2, 4, and 6 hours post-dose. Day 7: predose; 1, 2, 4, and 6 hours post-dose
Population: Due to the small sample size (n=2), data cannot be reported without risking participant re-identification. Data are not being reported in order to protect participants' privacy.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

3. Primary Outcome: Phase 1: Cmin of Itacitinib When Administered With Corticosteroids
Description: Cmin was defined as the minimum observed plasma concentration.
Time Frame: Day 1: 1, 2, 4, and 6 hours post-dose. Day 7: predose; 1, 2, 4, and 6 hours post-dose
Population: as for outcome 2
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

4. Primary Outcome: Phase 1: Tmax of Itacitinib When Administered With Corticosteroids
Description: Tmax was defined as the time to the maximum concentration.
Time Frame: Day 1: 1, 2, 4, and 6 hours post-dose. Day 7: predose; 1, 2, 4, and 6 hours post-dose
Population: as for outcome 2
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

5. Primary Outcome: Phase 1: AUC of Itacitinib When Administered With Corticosteroids
Description: AUC was defined as the area under the plasma concentration-time curve.
Time Frame: Day 1: 1, 2, 4, and 6 hours post-dose. Day 7: predose; 1, 2, 4, and 6 hours post-dose
Population: as for outcome 2
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

6. Primary Outcome: Phase 1: Cl/F of Itacitinib When Administered With Corticosteroids
Description: Cl/F was defined as the apparent oral dose clearance.
Time Frame: Day 1: 1, 2, 4, and 6 hours post-dose. Day 7: predose; 1, 2, 4, and 6 hours post-dose
Population: as for outcome 2
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

7. Primary Outcome: Phase 2: Overall Response Rate up to Day 28
Description: Overall response rate was defined as the number of participants demonstrating a complete response (CR), a very good partial response (VGPR), or a partial response (PR).
Time Frame: up to Day 28
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase 2: Number of Participants With TEAEs
Description: A TEAE was defined as an AE that began or worsened from Baseline after the first administration of study drug.
Time Frame: up to 12 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase 2: Cmax of Itacitinib When Administered With Corticosteroids
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Day 7: predose; 1, 2, and 4 hours post-dose
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase 2: Cmin of Itacitinib When Administered With Corticosteroids
Description: Cmin was defined as the minimum observed plasma concentration.
Time Frame: Day 7: predose; 1, 2, and 4 hours post-dose
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase 2: Tmax of Itacitinib When Administered With Corticosteroids
Description: Tmax was defined as the time to the maximum concentration.
Time Frame: Day 7: predose; 1, 2, and 4 hours post-dose
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase 2: AUC of Itacitinib When Administered With Corticosteroids
Description: AUC was defined as the area under the plasma concentration-time curve.
Time Frame: Day 7: predose; 1, 2, and 4 hours post-dose
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 2: Cl/F of Itacitinib When Administered With Corticosteroids
Description: Cl/F was defined as the apparent oral dose clearance.
Time Frame: Day 7: predose; 1, 2, and 4 hours post-dose
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 2: Overall Response Rate up to 100 Days
Description: Overall response rate was defined as the number of participants demonstrating a CR, a VGPR, or a PR.
Time Frame: up to 100 days
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 1: Overall Response Rate
Description: Overall response rate was defined as the number of participants demonstrating a CR, a VGPR, or a PR.
Time Frame: up to Day 28
Population: The study was terminated before participants reached Day 28, the time point for analysis.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase 2: Non Relapse Mortality
Description: Non relapse mortality was defined as the number of participants who died due to causes other than underlying hematologic disorders relapse.
Time Frame: up to 24 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase 2: Duration of Response
Description: Duration of response was defined as the time of the onset of response to the loss of response.
Time Frame: up to approximately 12 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

18. Secondary Outcome: Phase 2: Time to Response
Description: Time to response was defined as the interval from treatment initiation to the first response.
Time Frame: up to approximately 12 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

19. Secondary Outcome: Phase 2: Relapse Rate of Malignant and Nonmalignant Disorders
Description: Relapse rate was defined as the number of participants whose underlying disease relapsed.
Time Frame: up to approximately 12 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

20. Secondary Outcome: Phase 2: Malignant and Nonmalignant Disorders Relapse-related Mortality Rate
Description: Mortality rate was defined as the number of participants whose underlying hematologic disorder relapsed and had a fatal outcome.
Time Frame: up to approximately 12 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

21. Secondary Outcome: Phase 2: Failure-free Survival
Description: Failure-free survival was defined as the number of participants who were still alive, had not relapsed, had not required additional therapy for acute graft-versus-host disease (aGVHD), and had not demonstrated signs or symptoms of chronic GVHD.
Time Frame: up to 6 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

22. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival was defined as the interval from study enrollment to death due to any cause.
Time Frame: up to approximately 12 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

23. Secondary Outcome: Phase 2: Incidence Rate of Secondary Graft Failure
Description: Analysis was to be conducted to assess the number of participants experiencing secondary graft failure.
Time Frame: up to approximately 12 months
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

24. Secondary Outcome: Phase 2: Average Corticosteroid Use
Description: The average number of participants who discontinued corticosteroids was to be assessed.
Time Frame: up to 180 days
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

25. Secondary Outcome: Phase 2: Cumulative Corticosteroid Dose
Description: The number of participants with various cumulative corticosteroid doses was assessed.
Time Frame: up to 180 days
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

26. Secondary Outcome: Phase 2: Number of Participants Who Discontinued Corticosteroids
Description: The number of participants who discontinued corticosteroids was assessed.
Time Frame: up to 100 days
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

27. Secondary Outcome: Phase 2: Number of Participants Who Discontinued Immunosuppressive Medication
Description: The number of participants who discontinued immunosuppressive medication was assessed.
Time Frame: up to 100 days
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

28. Secondary Outcome: Phase 2: Number of Participants With aGVHD Flares
Description: The number of participants who experienced aGVHD flares requiring treatment was assessed.
Time Frame: up to 100 Days
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

29. Secondary Outcome: Phase 2: Number of Participants With Chronic Graft-versus-host Disease (cGVHD)
Description: The number of participants with a diagnosis of any cGVHD, including mild, moderate, severe, was assessed.
Time Frame: up to 365 days
Population: No participants enrolled in Phase 2 due to early termination of the study.
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 45 days
Arm/Group | Cohort 1 : Itacitinib + Corticosteroids
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 : Itacitinib + Corticosteroids (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Parvovirus infection (Infections and infestations) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 : Itacitinib + Corticosteroids (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03721965/Prot_SAP_000.pdf